CLINICAL TRIAL: NCT07294625
Title: A Clinical Study to Evaluate the Safety, Tolerability, and Efficacy of the LVIVO-TaVec200 Product in the Treatment of Relapsed/Refractory Multiple Myeloma
Brief Title: A Clinical Study to Evaluate LVIVO-TaVec200 for the Treatment of Relapsed/Refractory Multiple Myeloma
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Collaborators: Nanjing Legend Biotech Co. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LB2503-0001
Record Dates: First submitted 2025-12-08; First posted 2025-12-19 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Multiple Myeloma
Keywords: Relapsed/Refractory multiple myeloma
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- LVIVO-TaVec200 product (Experimental): Each subject will be given a single-dose LVIVO-TaVec200 product infusion at each dose level
  Interventions: Biological: LVIVO-TaVec200 product

INTERVENTIONS:
Biological: LVIVO-TaVec200 product — Prior to infusion of the LVIVO-TaVec200 product, subjects will receive bridging therapy if needed.

SUMMARY:
This is a prospective, single-arm, open-label dose-escalation clinical study to evaluate LVIVO-TaVec200 in the treatment of relapsed/refractory multiple myeloma.

DETAILED DESCRIPTION:
This is a prospective, single-arm, open-label dose-escalation and dose-expansion study, designed to evaluate the safety, tolerability, anti-tumor efficacy profile, and pharmacokinetic characteristics of the LVIVO-TaVec200 in subjects with relapsed/refractory multiple myeloma who have failed at least 3 lines of prior standard therapies. The subject who meet the defined eligibility criteria will be enrolled with a core study period of approximately 2 years, including the screening, bridging therapy(if needed), treatment, and follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects voluntarily participate in clinical studies; Fully informed of this study and signed informed consent; Informed consent form must be obtained prior to initiation of any study-related tests or procedures that are not part of the standard treatment for the subject's disease; Good compliance and cooperation with follow-up.
2. Age ≥ 18 years.
3. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
4. Has measurable lesions
5. Relapsed and/or refractory multiple myeloma
6. Life expectancy≥ 3 months
7. Clinical laboratory values meet screening visit criteria
8. Adequate organ function.

Exclusion Criteria:

1. Prior antitumor therapy with insufficient washout period ;
2. Prior treatment targeting GPRC5D;
3. Patients who are positive for hepatitis B surface antigen (HBsAg), hepatitis B virus deoxyribonucleic acid (HBV DNA), hepatitis C antibody (HCV-Ab), hepatitis C virus ribonucleic acid (HCV RNA), and human immunodeficiency virus antibody (HIV-Ab).
4. Known life-threatening allergic reaction, hypersensitivity reaction, or intolerance to study drug excipients and related excipients, including but not limited to DMSO; or those with a history of severe allergic reactions in the past (such as hypersensitivity reactions, or those with severe immune-related reactions such as the need for glucocorticoids to prevent anaphylaxis as assessed by the investigator).
5. Any condition deemed by the investigator as rendering the subject unsuitable for participation in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2025-12-10 (Estimated); Primary Completion 2027-03-31 (Estimated); Study Completion 2029-03-31 (Estimated)

PRIMARY OUTCOMES:
Incidence, severity and type of TEAEs (Treatment-emergent Adverse Events) | Through study completion, an average of 2 years after LVIVO-TaVec200 infusion (Day 1)
  An adverse event is any untoward medical event that occurs in a participant administered an investigational product, and it does not necessarily indicate only events with clear causal relationship with the relevant investigational product.
Pharmacokinetics in peripheral blood | Through study completion, an average of 2 years after LVIVO-TaVec200 infusion (Day 1)
  CAR positive T cells and CAR transgene percentage of in peripheral blood after LVIVO-TaVec200 infusion
Pharmacokinetics in bone marrow | Through study completion, an average of 2 years after LVIVO-TaVec200 infusion (Day 1)
  CAR positive T cells and CAR transgene percentage of in bone marrow after LVIVO-TaVec200 infusion
The recommended Phase II dose (RP2D) for this cell | 30 days after LVIVO-TaVec200 infusion
  RP2D established through BF-BOIN design and the DLTs occurring following LVIVO-TaVec200 infusion

CONTACTS AND LOCATIONS:
Locations (5):
- China (5):
  - Henan Cancer Hospital, Zhengzhou, Henan
  - The First Affiliated Hospital with Nanjing Medical University, Nanjing, Jiangsu
  - The Affiliated Hospital of XUZHOU Medical University, Xuzhou, Jiangsu
  - Ruijin Hospital Affiliated to Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality
  - The Second Affiliated Hospital of Xi'an Jiaotong University, Xi’an, Shanxi

IPD SHARING:
Plan to Share IPD: No